CLINICAL TRIAL: NCT05412719
Title: The Effect Of Finger Pupiling On Pain And Physiological Parameters During Urinary Culture With Urinary Catheter in İnfants
Brief Title: The Effect Of Finger Pupiling On Pain And Physiological Parameters in İnfants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Duygu Cicek, duygu çiçek, Okan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021/210
Record Dates: First submitted 2022-05-13; First posted 2022-06-09 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-05

CONDITIONS: Pain
Keywords: pain, infants
MeSH Terms: conditions — Pain | interventions — Urinary Catheterization

STUDY DESIGN:
Intervention Model Description: Randomized Controlled two groups (control group and intervention group)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Experimental): . Before the procedure, the baby's pulse, blood pressure, SpO2, respiratory rate were checked by an observing nurse and recorded on the Baby Monitoring Form.
  * An observer nurse will assist the doctor at the beginning of the procedure, and then the baby's upper legs are kept stable in order to maintain the stability of the baby and ensure that the doctor can see the urethral opening. The other observer nurse evaluated the respiratory rate of the baby during the procedure and recorded it in the Infant Follow-up Form after the procedure was completed.
  * During the procedure, the baby was evaluated by both observer nurses according to the FLAAC pain scale.
  * No pharmacological or non-pharmacological interventions were made for the baby's pain during the procedure.
  Interventions: Behavioral: THE EFFECT OF FINGER PUPPET MANIPULATION ON PAİN AND PHYSİOLOGıCAL PARAMETERS DURING URINARY CULTURE WITH URINARY CATHETERIZATION IN INFANTS
- intervention group (Experimental): Before the procedure, the baby's heart rate, blood pressure, spo2, respiratory rate, FLACC were recorded, 5 minutes before the procedure, the finger puppet was started to be played by singing the red fish song, the baby's pulse, spo2, respiratory rate and FLACC scale were recorded during the procedure, 5 minutes after the procedure Playing more finger puppetry Evaluation of the baby's pulse, blood pressure, spo2, respiratory rate and FLAAC immediately after the procedure and five minutes later
  Interventions: Behavioral: THE EFFECT OF FINGER PUPPET MANIPULATION ON PAİN AND PHYSİOLOGıCAL PARAMETERS DURING URINARY CULTURE WITH URINARY CATHETERIZATION IN INFANTS

INTERVENTIONS:
Behavioral: THE EFFECT OF FINGER PUPPET MANIPULATION ON PAİN AND PHYSİOLOGıCAL PARAMETERS DURING URINARY CULTURE WITH URINARY CATHETERIZATION IN INFANTS — the effect of finger puppet manipulation on pain and physiological parameters during urinary culture with urinary catheterization
  Other Names: the effect of finger puppet manipulation on pain and physiological parameters during urinary culture with urinary catheterization

SUMMARY:
. In this determined, it was carried out to determine the effect of finger puppet play on pain and physiological parameters during urine culture with urinary catheter in infants.

Research Hypotheses and Variables H0: There is no difference between the pain levels of babies who were manipulated with finger puppets during urine culture sampling with urinary catheter compared to babies in the control group.

H1: Babies whose finger puppet is played during urine culture sampling with urinary catheter have low pain levels.

H2: Physiological parameters of babies who are played with finger puppets during urine culture sample collection with urinary catheter are positively affected.

DETAILED DESCRIPTION:
The research was designed as a randomizer controlled experimental study to determine the effect of finger puppet manipulation on pain and physiological catheter parameters during urinary culture with urinary catheterization in 2-12 month old infants. This Research was conducted in pediatric emergency department of SBU Zeynep Kamil Women's and Children's Diseases Training and Research Hospital between Feb.2021-Feb.2022. "Infant follow-up form" and "FLAAC pain scale" were used to collect data. The data obtained from the research were analyzed with appropriate statistical tests in the SPSS 22.0 package program.

Research Hypotheses and Variables H0: There is no difference between the pain levels of babies who were manipulated with finger puppets during urine culture sampling with urinary catheter compared to babies in the control group.

H1: Babies whose finger puppet is played during urine culture sampling with urinary catheter have low pain levels.

H2: Physiological parameters of babies who are played with finger puppets during urine culture sample collection with urinary catheter are positively affected.

Dependent Variables: Infants' physiological parameters (Pulse, Blood pressure, Respiration, SpO2) and Infant Follow-up Form, FLACC pain scale.

Independent Variables: Baby's age, gender. Sampling inclusion criteria

* The baby is between 2 and 12 months
* Suspicion/diagnosis of urinary tract infection being followed
* The baby/child does not have a vision or hearing problem (sight-hearing screening tests have been completed)
* Not taking drugs containing analgesics in the last 4 hours before the procedure
* Parents' willingness to participate in the research
* It has been determined as the appropriate cognitive level and motor development of infants/children.

Exclusion criteria

* Mentally or neurologically handicapped
* Having a life-threatening illness
* Babies who failed the procedure, took longer than 3 minutes and needed to be repeated were excluded from the sample.

Data were collected using the Baby Monitoring Form, monitor and sphygmomanometer Infant Follow-up Form: After the written Informed Consent Form (Appendix-1) was obtained from the parents of the infants who met the conditions for participation in the study, stating that they volunteered to participate in the study, the data were collected by the researcher, questioning the age, gender, current complaint, whether the procedure was performed before, and his reaction to the procedure. 7 questions were collected with the Infant Follow-up Form, which included physiological parameters (pulse, blood pressure, SpO2, respiratory rate) and the FLACC pain scale (Appendix-2).

FLACC Pain Scale: It is an observational behavioral pain scale used in infants and children who cannot express their pain verbally. It is used for babies and children aged 2 months to 7 years. It consists of five categories that measure the baby's facial expression, leg movements, activity, crying, and comfortability. Each of the categories is scored between 0-2, and a total score of 0-10 is obtained, and an increase in the score indicates that the pain also increases. The total score according to the scoring system made after the observation; 0: comfortable, calm, comfortable, 1-3: mildly uncomfortable or mild pain, 4-6: moderate pain, 7-10: significant severe discomfort or significant severe pain, or both. The FLACC pain scale was evaluated independently by two different observers.

Bedside Monitor Device: A COVIDIEN Nellcor brand monitor was used to measure the patient's pulse and SpO2.

Blood pressure monitor: A Unitest brand digital sphygmomanometer with a cuff compatible with the baby was used.

Finger Puppet: Fish-shaped finger puppet made of red fabric is used. Families of infants who were admitted to the emergency department and followed up with the diagnosis/suspect of urinary tract infection were informed about the study by face-to-face interview technique, and the informed consent form prepared by the researcher was read and permission was obtained. Out of 80 infants aged 2-12 months, 40 infants (intervention group: finger puppet group) and 40 infants (control group) were divided into two groups. In order to assign the babies to the groups randomly, between the dates of the study, the babies who would be treated on odd number days of the calendar formed the group to be treated with finger puppets, and the baby who was treated on even number days constituted the control group.

First of all, the procedure to be done was explained to the family. Written and verbal consent was obtained after giving information about the study. During the procedure, the family was informed that only the mother, the physician performing the procedure, the researcher and the observer nurses would be present in the room.

Urine culture with the urinary catheterization method is a procedure performed by the physician under sterile conditions for approximately 1-3 minutes. A finger puppet was played by the researcher nurse in the intervention group by singing the red fish song in order to manage the pain during the invasive procedure and to distract the baby's attention.

Initiative Group (Finger Puppet Played Group)

* The baby to be treated was taken to the intervention room by the research nurse.
* Before the procedure, the baby's pulse, blood pressure, SpO2, respiratory rate will be checked by an observing nurse and recorded on the Baby Monitoring Form.
* Before the procedure, the infant was recorded in the Infant Follow-up Form by evaluating the FLAAC pain scale independently by both observer nurses.
* 5 minutes before the start of the procedure, a red fish-shaped finger puppet was started to be played by the research nurse by singing the red fish song from a distance of approximately 20-30 cm.
* An observer nurse will assist the physician at the beginning of the procedure, and then gently hold the infant by the upper legs to maintain the stability of the infant and ensure that the physician can see the urethral opening. The other observer nurse evaluated the respiratory rate of the baby during the procedure and recorded it in the Infant Follow-up Form after the procedure was completed.
* During the procedure, the baby was independently evaluated according to the FLAAC pain scale by both observer nurses.
* The research nurse will continue to play finger puppets for 5 more minutes after the end of the procedure, and the puppet play was terminated after 5 minutes.
* Immediately after the procedure and five minutes later, the baby's pulse, blood pressure, SpO2, respiratory rate will be checked and the baby's pain was evaluated by both observer nurses according to the FLAAC pain scale, recorded in the Baby Monitoring Form, and then the baby was delivered to the family.
* During the procedure, no pharmacological or non-pharmacological interventions were made for the baby's pain, and no attempts were made to distract the baby's attention except finger puppets

Control group:

* The baby to be treated was taken to the intervention room by the research nurse.
* Before the procedure, the baby's pulse, blood pressure, SpO2, respiratory rate were checked by an observing nurse and recorded on the Baby Monitoring Form.
* An observer nurse will assist the doctor at the beginning of the procedure, and then the baby's upper legs are kept stable in order to maintain the stability of the baby and ensure that the doctor can see the urethral opening. The other observer nurse evaluated the respiratory rate of the baby during the procedure and recorded it in the Infant Follow-up Form after the procedure was completed.
* During the procedure, the baby was evaluated by both observer nurses according to the FLAAC pain scale.
* No pharmacological or non-pharmacological interventions were made for the baby's pain during the procedure.
* Immediately after the procedure and 5 minutes later, the baby's pulse, blood pressure, SpO2, respiratory rate were checked and recorded, and both observer nurses independently evaluated the baby's pain according to the FLAAC Pain Scale and recorded it in the Baby Monitoring Form, and then the baby was delivered to the family.

The quantitative data obtained in the research will be analyzed in the computer environment after data entry is made in the SPSS 21.0 package program. Number, percentage, mean and standard deviation were used as descriptive statistical methods in the evaluation of the data. Before the data analysis, the normality test was performed to test the suitability for the parametric test methods. In order to test the normal distribution condition, Kolmogorov-Smirnov Z test was applied. Chi-square and fisherexact tests were applied to determine the homogeneity of the groups. Whether there is a statistical difference between the groups, repeated measurements; Pairwise comparison was evaluated with Independent group t-test. The findings were evaluated at 95% confidence interval and 5% significance level. It was stated that there was a significant difference between the groups when p<0.05, and there was no significant difference in case of p>0.05.

Before starting the research, ethics committee approval from the Research Zeynep Kamil Gynecology and Pediatrics Training and Research Hospital Ethics Committee , Master's Thesis Work Permit from Istanbul Provincial Health Directorate , translation of FLACC Pain Scale into Turkish was required. necessary permissions were obtained.

After the parents of the infants included in the study were informed about the study, their written consent was obtained with the "Informed Voluntary Consent Form" .

ELIGIBILITY:
Inclusion Criteria:

* The baby is between 2 and 12 months

  * Suspicion/diagnosis of urinary tract infection being followed
  * The baby/child does not have a vision or hearing problem (sight-hearing screening tests have been completed)
  * Not taking drugs containing analgesics in the last 4 hours before the procedure
  * Parents' willingness to participate in the research
  * It has been determined as the appropriate cognitive level and motor development of infants/children

Exclusion Criteria:

Mentally or neurologically handicapped

* Having a life-threatening illness
* Babies who failed the procedure, took longer than 3 minutes and needed to be repeated were excluded from the sample

Ages: 2 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
pain score | before urinary catheter intervention(5 minutes ago)
  It is used for babies and children aged 2 months to 7 years. It consists of five categories that measure the baby's facial expression, leg movements, activity, crying, and comfortability. A total of 0-10 points are obtained in the scale, where each of the categories is scored between 0-2, and the increase in the score indicates that the pain also increases. According to the scoring system made after the observation, the total score is 0: the child is comfortable, calm, comfortable, 1-3: slightly uncomfortable. or mild pain, 4-6: moderate pain, 7-10: significant severe discomfort or significant severe pain, or both.
pain score | urinary catheter attempt sequence (0th minute)
  It is used for babies and children aged 2 months to 7 years. It consists of five categories that measure the baby's facial expression, leg movements, activity, crying, and comfortability. A total of 0-10 points are obtained in the scale, where each of the categories is scored between 0-2, and the increase in the score indicates that the pain also increases. According to the scoring system made after the observation, the total score is 0: the child is comfortable, calm, comfortable, 1-3: slightly uncomfortable. or mild pain, 4-6: moderate pain, 7-10: significant severe discomfort or significant severe pain, or both.
pain score | immediately after urinary catheter interventioan (0th minute)
  It is used for babies and children aged 2 months to 7 years. It consists of five categories that measure the baby's facial expression, leg movements, activity, crying, and comfortability. A total of 0-10 points are obtained in the scale, where each of the categories is scored between 0-2, and the increase in the score indicates that the pain also increases. According to the scoring system made after the observation, the total score is 0: the child is comfortable, calm, comfortable, 1-3: slightly uncomfortable. or mild pain, 4-6: moderate pain, 7-10: significant severe discomfort or significant severe pain, or both.
pain score | 5 minutes after urinary catheterization
  It is used for babies and children aged 2 months to 7 years. It consists of five categories that measure the baby's facial expression, leg movements, activity, crying, and comfortability. A total of 0-10 points are obtained in the scale, where each of the categories is scored between 0-2, and the increase in the score indicates that the pain also increases. According to the scoring system made after the observation, the total score is 0: the child is comfortable, calm, comfortable, 1-3: slightly uncomfortable. or mild pain, 4-6: moderate pain, 7-10: significant severe discomfort or significant severe pain, or both.
SPO2 vital signs | before urinary catheter intervention(5 minutes ago)
  SPO2 (%) were evaluated
SPO2 vital signs | urinary catheter attempt sequence (0th minute)
  SPO2 (%) were evaluated
SPO2 vital signs | immediately after urinary catheter interventioan (0th minute)
  SPO2 (%) were evaluated
SPO2 vital signs | 5 minutes after urinary catheterization
  SPO2 (%) were evaluated
blood pressure vital signs | before urinary catheter intervention(5 minutes ago)
  blood pressure (mmHg) were evaluated
blood pressure vital signs | immediately after urinary catheter interventioan (0th minute)
  blood pressure (mmHg) were evaluated
blood pressure vital signs | 5 minutes after urinary catheterization
  blood pressure (mmHg) were evaluated
heart rate vital signs | before urinary catheter intervention(5 minutes ago)
  heart rate (beats/minute) were evaluated
heart rate vital signs | urinary catheter attempt sequence (0th minute)
  heart rate (beats/minute) were evaluated
heart rate vital signs | immediately after urinary catheter interventioan (0th minute)
  heart rate (beats/minute) were evaluated
heart rate vital signs | 5 minutes after urinary catheterization
  heart rate (beats/minute) were evaluated
respiratory rate vital signs | before urinary catheter intervention(5 minutes ago)
  respiratory rate (beats/minute) were evaluated
respiratory rate vital signs | urinary catheter attempt sequence (0th minute)
  respiratory rate (beats/minute) were evaluated
respiratory rate vital signs | immediately after urinary catheter interventioan (0th minute)
  respiratory rate (beats/minute) were evaluated
respiratory rate vital signs | 5 minutes after urinary catheterization
  respiratory rate (beats/minute) were evaluated

CONTACTS AND LOCATIONS:
Locations (1):
- Okan University, Istanbul, Tuzla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No